CLINICAL TRIAL: NCT00784784
Title: A Pilot Study for a Randomized Controlled Trial to Compare Trivalent Split Virus Influenza Vaccine to Seasonal Antiviral Prophylaxis in Healthcare and Other Healthy Adults: Assessment of Zanamivir Versus Vaccine (Stop-Flu-2)
Brief Title: Zanamivir Versus Trivalent Split Virus Influenza Vaccine
Acronym: Stop-Flu-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Dr. Allison McGeer/Director, Infection Control, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-0189-A; CRT113936 (Other Grant/Funding Number: GSK)
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Influenza
Keywords: antiviral drugs; influenza vaccines
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Zanamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccine (Experimental): Influenza vaccine, using Fluviral trivalent split virus vaccine
  Interventions: Biological: Fluviral
- Antiviral prophylaxis (Experimental): Zanamivir antiviral prophylaxis
  Interventions: Drug: Zanamivir

INTERVENTIONS:
Biological: Fluviral — One dose
  Arms: Influenza vaccine
Drug: Zanamivir — 10 mg, OD, for duration of influenza season (10-23 weeks)
  Other Names: Relenza
  Arms: Antiviral prophylaxis

SUMMARY:
This unblinded pilot study is intended to assess the feasibility of a larger double-blind, randomized control trial. For the larger trial the investigators are interested in understanding the relative benefits of vaccine and antiviral prophylaxis, the risk factors for influenza infection in healthy adults, and in assessing the safety and tolerability of seasonal antiviral prophylaxis in healthcare workers.

The pilot study will be assessing the rate of infection with influenza and the rate of adherence to long-term zanamivir in 60 healthy volunteers.

DETAILED DESCRIPTION:
Several studies have demonstrated that zanamivir and oseltamivir are effective in preventing influenza infection and illness when used either as prophylaxis after exposure to a household contact with influenza or when taken for several weeks at the height of influenza activity in the general community. However, the longest duration of prophylaxis with neuraminidase inhibitors in two clinical trials, to date, has been six weeks.

Antiviral medication will likely have an important role in the response to the next influenza pandemic. Additionally, there may be indications for use during seasons when the major infecting strain of influenza in not one whose antigen is well covered by the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* 18-69 years old as of 01/Nov/2008
* have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry
* available for follow-up during the study period
* if a women of child-bearing years, must meet criteria to prevent pregnancy

Exclusion Criteria:

* allergy to any component of influenza vaccine or zanamivir
* previous serious adverse event associated with influenza vaccination
* receipt of influenza vaccine between 01/Mar/2008 and start of study
* previous adverse event associated with the use of antiviral medications
* expecting to be unable to take zanamivir for more than 72 hours during study period
* planning to spend more than 2 consecutive weeks outside Canada or more than 100 km from the study site during study period
* pregnant, or planning to become pregnant, during study period
* breastfeeding, or planning to breastfeed, a child under 12 months of age during study period
* receipt of immunoglobulin within six months of study entry
* immunocompromising condition or therapy that would be expected to reduce the efficacy of vaccination
* plans to receive cytotoxic or radiation therapy during study period
* history of cardiovascular or pulmonary disease that has required hospital admission within the past year
* history of asthma or other chronic respiratory disease
* participating in a trial that will result in the receipt of an investigational medication during the period that zanamivir may be taken (15/Nov/2008 to 30/Apr/2009)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison McGeer, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 5th to November 19th, 2008 in Toronto, Ontario Canada. Most subjects were healthcare workers employed at a 470-bed acute care facility.
Groups:
- Antiviral Prophylaxis: Zanamivir, 10mg once daily during period of influenza activity, as prophylaxis
Period: Overall Study
Arm/Group | Influenza Vaccine | Antiviral Prophylaxis
Started | 22 | 42
Completed | 20 | 40
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine | Antiviral Prophylaxis | Total
Number analyzed (Participants) | 22 | 42 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 42 | 64
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10) | 40 (10) | 40 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 27 | 44
  Male | 5 | 15 | 20
Region of Enrollment [Number; unit: participants]
  Canada | 22 | 42 | 64

OUTCOME MEASURES:

1. Secondary Outcome: Number of Subjects Adhering to Long-term Zanamivir Prophylaxis
Description: Number of subjects taking 80% or more doses per week of zanamivir (10 mg once daily), as influenza prophylaxis, for 13 weeks or longer (as measured by weekly diary and dose counts at study visits).
Time Frame: 5 months
Population: ITT
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Influenza Vaccine | Antiviral Prophylaxis
Number analyzed (Participants) | 0 | 40
participants |  | 34 [29 to 37]

2. Primary Outcome: Number of Laboratory Confirmed Influenza Infections
Description: Four-fold increase in antibody titer 2 weeks post injection and end of study or positive laboratory test for influenza during study (polymerase chain reaction [PCR] or culture)
Time Frame: 6 months
Population: intention to treat
Measure: Number; unit: infections
Arm/Group | Influenza Vaccine | Antiviral Prophylaxis
Number analyzed (Participants) | 20 | 40
infections | 2 | 1
Statistical Analysis 1: Comparison: Influenza Vaccine vs Antiviral Prophylaxis; That in a year with mismatch between influenza vaccine antigen and infecting H3N2 strain, seasonal (10-13 weeks) antiviral prophylaxis in adults will provide better protection from symptomatic influenza infection than trivalent inactivated split virus influenza vaccine; Test type: Superiority or Other; p = 0.25, Fisher Exact; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.01 to 4.8]

ADVERSE EVENTS:
Time Frame: 7 months
Description: Solicited and unsolicited adverse event reporting
Arm/Group | Influenza Vaccine | Antiviral Prophylaxis
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/40
Other Adverse Events (participants affected / at risk) | 0/22 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza Vaccine (N=20) | Antiviral Prophylaxis (N=40)
Broken bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Pilot study: Limited number of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No